CLINICAL TRIAL: NCT05198154
Title: A Multicenter, Prospective Clinical Study of Circulating Tumor DNA Analysis to Monitor the Risk of Progression After Long-term Benefit to First-line Immunotherapy in Patients With Advanced NSCLC (CR1STAL)
Brief Title: ctDNA Analysis to Monitor the Risk of Progression After First-line Immunotherapy in Patients With Advanced NSCLC
Acronym: CR1STAL
Status: Recruiting | Type: Observational
Sponsor: Fang Wu (Other)
Collaborators: Sun Yat-sen University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Fujian Cancer Hospital (Other Government); Third Affiliated Hospital of Third Military Medical University (Other); Xiangya Hospital of Central South University (Other); Qinghai Province Tumor Hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhejiang Provincial People's Hospital (Other); Hunan Province Tumor Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Cancer Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Inner Mongolia People's Hospital (Other); Guizhou Provincial People's Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Yueyang Central Hospital (Other); ZhuZhou Central Hospital (Other); Zhangjiajie Affiliated Hospital of Hunan Normal University (Unknown); Loudi Central Hospital (Other); Chang Sha First Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Fang Wu, Associate Professor, Second Xiangya Hospital of Central South University
Organization: Second Xiangya Hospital of Central South University (Other)
Other Study IDs: XYEYY20211024
Record Dates: First submitted 2022-01-01; First posted 2022-01-20 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-02

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma
Keywords: ctDNA; advanced lung cancer; first-line immunotherapy; the risk of progression; minimal residual disease (MRD); long-term benefit
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma cell free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Advanced NSCLC patients with long-term benefit after first-line immunotherapy (Tumor-informed group): The ctDNA detection will be performed using a tumor-informed analysis approach. This method requires the availability of tumor tissue samples or a fixed-panel next-generation sequencing (NGS) test.
  Interventions: Diagnostic Test: ctDNA detection
- Advanced NSCLC patients with long-term benefit after first-line immunotherapy (Tumor-agnostic group): The ctDNA detection will be performed using a tumor-agnostic analysis. This method does not require tumor tissue samples or an NGS testing panel, or in cases where tissue samples are available but fail to meet quality control standards.
  Interventions: Diagnostic Test: ctDNA detection

INTERVENTIONS:
Diagnostic Test: ctDNA detection — High-depth sequencing method is used to detecting ctDNA.

SUMMARY:
This study aims to explore the correlation of circulating tumor DNA(ctDNA) and the risk of progression in patients with advanced NSCLC who have long-term benefit from first-line immunotherapy (PFS 12 months)

DETAILED DESCRIPTION:
Evidence suggests that circulating tumor DNA (ctDNA) analysis can noninvasively identify minimal residual disease (MRD) in clinical oncology. The researches will be sharply increased about ctDNA potential clinical application in the near future. In the early stage of NSCLC, ctDNA has been indicated to identify those at high risk of recurrence after radical surgery. And this study will focus on those patients with advanced NSCLC who have long-term benefit from first-line immunotherapy (PFS 12 months). 10ml plasma will be collected every three months until disease progression to interrogate ctDNA by high-depth panel sequencing, exploring its prediction value about the risk of progression. Meanwhile, the investigators would like to explore the lead time of detectable ctDNA before regular imaging finding.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Advanced non-small cell lung cancer (stage IIIB-IV), pathological types limited to squamous cell carcinoma or non-squamous cell carcinoma, driver gene mutations (EGFR/ALK/ROS1) were negative
* General condition: ECOG score 0 or 1
* First-line monotherapy or combination immunotherapy
* The long-term benefit of immunotherapy was defined as PFS=12months
* Tumor tissue samples can be obtained at the time of enrollment, and at least 5 ~ 10 sections can be generated, and the pathological report indicates that the overall tumor content is not less than 10% or NGS testing with a fixed-panel is available; or no tumor tissue is available.
* At least one measurable lesion (except patients with CR after first-line treatment) can be evaluated according to RECIST1.1 standard.
* Have self-awareness, be able to understand the research scheme and voluntarily participate in the study, and can sign the informed consent form
* Have good compliance, be able to cooperate with the collection of specimens from each node and provide corresponding clinical information.

Exclusion Criteria:

* Serious primary diseases of the heart, liver and kidney
* Other malignant tumors within 3 years prior to diagnosis of NSCLC
* Women in pregnancy and lactation
* The active stage of human immunodeficiency virus (HIV) infection
* Patients with active systemic infection, pneumonia, tuberculosis, pericarditis
* Patients who cannot understand the content of the experiment and cannot cooperate and refuse to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically confirmed advanced NSCLC patients with long-term benefit after first-line immunotherapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  The duration from study enrollment to disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
The correlation of ctDNA and risk of progression | 3 years
  The correlation of ctDNA and risk of progression during the erolled observation process
Lead time | 3 years
  Lead time defined as the interval between ctDNA detection and imaging of progression.
Incidence of adverse events | 3 years
  the incidence of adverse events during the whole observation time
Overall survival (OS) | 3 years
  Overall survival (OS) defined as the duration from study enrollment until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.

OTHER OUTCOMES:
Objective response rate (ORR) | 3 years
  ORR is defined as the proportion of study participants who achieve complete response (CR) or partial response (PR) among the total study participants.
Factors influencing ctDNA detection | 3 years
  Analyze the factors affecting ctDNA shedding and non-shedding.
Differences between ctDNA MRD and other peripheral blood biomarkers. | 3 years
  Differences between ctDNA MRD and other peripheral blood biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department，Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided